CLINICAL TRIAL: NCT04434573
Title: Asymptomatic Abdominal Wall and Incisional Hernias: Is Therapeutic Decision Consensual An International Survey
Brief Title: Consensus in Surgical Community for Asymptomatic Abdominal Wall and Incisional Hernias
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 20_213
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Study of Practices of Surgeons on Surgical Management of Asymptomatic Hernias; Comparison With International Recommendations
MeSH Terms: interventions — Observational Studies as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- french-speaking digestive surgeons: french-speaking digestive surgeons are visceral and digestive surgeons that have a general surgical activity too. They can have or not an expertise on hernia pathology. They are questioned by survey on decisions about different patient asymptomatic hernia clinical situations.
  Interventions: Other: Observation study

INTERVENTIONS:
Other: Observation study — French-speaking digestive surgeons are invited to respond to an online survey consisting of 13 common clinical situations concerning primary or asymptomatic incisional hernia pathology where a therapeutic decision is requested.

SUMMARY:
Hernia pathology is one of the leading causes of surgery worldwide. For asymptomatic patients, surgery remains questionable. Although there are new European recommendations, the practice of digestive surgeons regarding the management of asymptomatic hernias is unknown. The objective of this study was to evaluate the practices of a large population of digestive surgeons with asymptomatic hernia.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French-speaking surgeons
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
number and type of clinical cases for which a consensus, defined by an arbitrary value of 75% of surgeons with the same therapeutic attitude | The outcome measure is evaluated after 6 months during which the survey is online (from october 2016 to march 2017), time during which surgeons had access to answer it
  The survey consists of general questions about the surgeons' activity and then 13 clinical situations where a decision is requested. The clinical cases are developed by the authors of the study in order to solve the frequent problems with the treatment of hernias and incisional hernias

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, Île-de-France Region, France